CLINICAL TRIAL: NCT03978598
Title: Effect of Immediate Versus Standard Postpartum Insertion of the Contraceptive Implant on Breastfeeding Outcomes
Brief Title: Breastfeeding Etonogestrel Implant Study
Acronym: LACTO-Rod
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-049
Record Dates: First submitted 2019-05-24; First posted 2019-06-07 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immediate insertion group (Experimental): Immediate insertion in the first 24 hours after delivery ENG implant insertion Intervention.
  Interventions: Drug: Etonogestrel; Device: Nexplanon
- Standard Postpartum Insertion Group (Active Comparator): Insertion of the Etonogestrel implant 4-6 weeks postpartum Intervention.
  Interventions: Drug: Etonogestrel; Device: Nexplanon

INTERVENTIONS:
Drug: Etonogestrel — Immediate v. Standard insertion.
Device: Nexplanon — Implant.

SUMMARY:
The investigators are studying the effect of placing the etonogestrel implant (Nexplanon) in the first 24 hours after birth on breastfeeding. Women who wish to have an etonogestrel implant placed after their birth, wish to breastfeed, and are willing to participate in the study will be randomly assigned to either get the implant placed in the first 24 hours after delivery of the baby and placenta or 4-6 weeks later. The investigators do not believe there will be a difference in breastfeeding 8 weeks after delivery or time to lactogenesis between those who get the implant placed early or later.

DETAILED DESCRIPTION:
Counseling and provision of postpartum contraception is an integral component of comprehensive reproductive healthcare. A woman's preference for contraception is paramount; early initiation of postpartum contraception may assist in optimal birth spacing promoting the wellbeing of mother and baby. Equally important is the provision of appropriate support for breastfeeding. Exclusive breastfeeding for six months with continuation beyond one year of age is recommended by the American Academy of Pediatrics (AAP), American Academy of Family Physicians, American College of Obstetricians and Gynecologists (ACOG), and the World Health Organization (WHO).

The utilization of Long Acting Reversible Contraception (LARC's) has increased in the last decade. The etonogestrel (ENG) implant is one of the most effective LARC's and has become one of the methods used by many women in the postpartum period to prevent an unplanned pregnancy. The major advantage of immediate ENG implant insertion is the prompt initiation of a highly effective contraceptive method at a time that does not interfere with breastfeeding and the life changes and demands of motherhood.

Our long-term goal is to understand the impact of the ENG implant hormonal contraceptive, initiated early in the postpartum period, on breastfeeding. The central hypothesis is that breastfeeding continuation at eight weeks postpartum is not inferior in women in the immediate insertion group of the ENG implant than in those with standard insertion and that time to lactogenesis stage II is not more than 8 hours difference between the immediate insertion and standard insertion groups.

Primary:

Aim #1: To determine breastfeeding continuation rates at 8 weeks in both groups.

Aim #2: To determine the timing of lactogenesis in both groups

Secondary:

Aim #1: To assess breastfeeding continuation and exclusivity between the immediate versus the standard group. Aim #2: To compare postpartum factors associated with discontinuing breastfeeding between the immediate versus the standard group. Aim #3: To compare participant satisfaction with postpartum contraception counseling in women enrolled in the study and in those women who opted not to enroll in the study between the immediate versus the standard group. Aim #4: To compare postpartum mood as measured by EPDS score between the immediate versus the standard group. Aim #5: To compare postpartum sexual function as measured by Female Sexual Function Index (FSFI) score between the immediate versus the standard group. Aim #6: To compare the total number of days of postpartum bleeding in the immediate versus standard. Aim #7: To compare participant satisfaction with the timing of ENG implant insertion between the immediate versus the standard group

This proposal will support a non-inferiority RCT where participants will be randomly assigned to immediate insertion (first 24 hours after delivery) or delayed postpartum insertion (4-6 weeks postpartum). This project will provide needed evidence on breastfeeding impact of early postpartum initiation of the ENG implant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women or women who have delivered vaginally and by cesarean section within 22 hours (2-hour window will allow for implant insertion by 24 hours postpartum)
* Aged 13 and older
* English or Spanish speakers
* Deliver an infant at UNM Hospital at > 37 weeks gestational age
* Intend to breastfeed
* Desire the implant as a method for contraception
* Agree to randomization
* Must have a working phone (study questions to be answered through phone calls or accessed electronically by a link sent through email or text message)

Exclusion Criteria:

* Under age 13
* History of breast cancer (screen by past medical history)
* History of undiagnosed vaginal bleeding (screen by past medical history)
* Head trauma that affected pituitary function (screen by past medical history)
* Prolactin insufficiency (screen by past medical history)
* Previous lactation failure (defined as no lactation within 5 days postpartum)
* Any contraindication to lactation/implant use including diseases transmittable by breast milk (screen by past medical history)
* Liver dysfunction (screen by past medical history)
* Use of drugs that inhibit lactation (screen by medical history)
* Sensitivity to the components of the ENG implant (screen by past medical history)
* Contraindications to use the implant by the (US MEC) (screen by past medical history)
* Active labor
* Delivery at < 37 weeks gestational age

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Krashin@salud.unm.edu, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG committee opinion 736, Optimizing Postpartum Care. Washington, DC: American College of Obstetricians and Gynecologists. 2018 May; 131(5):140-150.
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] AAFP Releases Position Paper on Breastfeeding Am Fam Physician. 2015 Jan 1;91(1):56-57.
- [Background] ACOG Committee Opinion No. 756: Optimizing Support for Breastfeeding as Part of Obstetric Practice. Obstet Gynecol. 2018 Oct;132(4):e187-e196. doi: 10.1097/AOG.0000000000002890. PMID 30247365
- [Background] Infant and Young Child Feeding: Model Chapter for Textbooks for Medical Students and Allied Health Professionals. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK148965/ PMID 23905206
- [Background] CDC. 2018 Breastfeeding Report Card [Internet]. Centers for Disease Control and Prevention. 2018 [cited 2018 Nov 10]. Available from: https://www.cdc.gov/breastfeeding/data/reportcard.htm
- [Background] Chapman DJ, Perez-Escamilla R. Maternal perception of the onset of lactation is a valid, public health indicator of lactogenesis stage II. J Nutr. 2000 Dec;130(12):2972-80. doi: 10.1093/jn/130.12.2972. PMID 11110856
- [Background] Curtis KM, Tepper NK, Jatlaoui TC, Berry-Bibee E, Horton LG, Zapata LB, Simmons KB, Pagano HP, Jamieson DJ, Whiteman MK. U.S. Medical Eligibility Criteria for Contraceptive Use, 2016. MMWR Recomm Rep. 2016 Jul 29;65(3):1-103. doi: 10.15585/mmwr.rr6503a1. PMID 27467196
- [Background] Cunningham FG, Leveno KJ, Bloom SL, Dashe JS, Hoffman BL, Casey BM, et al. Contraception. In: Williams Obstetrics, 25e [Internet]. New York, NY: McGraw-Hill Education; 2018 [cited 2018 Nov 10].
- [Background] Turok DK, Leeman L, Sanders JN, Thaxton L, Eggebroten JL, Yonke N, Bullock H, Singh R, Gawron LM, Espey E. Immediate postpartum levonorgestrel intrauterine device insertion and breast-feeding outcomes: a noninferiority randomized controlled trial. Am J Obstet Gynecol. 2017 Dec;217(6):665.e1-665.e8. doi: 10.1016/j.ajog.2017.08.003. Epub 2017 Aug 23. PMID 28842126
- [Background] Sothornwit J, Werawatakul Y, Kaewrudee S, Lumbiganon P, Laopaiboon M. Immediate versus delayed postpartum insertion of contraceptive implant for contraception. Cochrane Database Syst Rev. 2017 Apr 22;4(4):CD011913. doi: 10.1002/14651858.CD011913.pub2. PMID 28432791
- [Background] Gurtcheff SE, Turok DK, Stoddard G, Murphy PA, Gibson M, Jones KP. Lactogenesis after early postpartum use of the contraceptive implant: a randomized controlled trial. Obstet Gynecol. 2011 May;117(5):1114-1121. doi: 10.1097/AOG.0b013e3182165ee8. PMID 21508750
- [Background] Phillips SJ, Tepper NK, Kapp N, Nanda K, Temmerman M, Curtis KM. Progestogen-only contraceptive use among breastfeeding women: a systematic review. Contraception. 2016 Sep;94(3):226-52. doi: 10.1016/j.contraception.2015.09.010. Epub 2015 Sep 26. PMID 26410174
- [Background] Bryant AG, Bauer AE, Stuart GS, Levi EE, Zerden ML, Danvers A, Garrett JM. Etonogestrel-Releasing Contraceptive Implant for Postpartum Adolescents: A Randomized Controlled Trial. J Pediatr Adolesc Gynecol. 2017 Jun;30(3):389-394. doi: 10.1016/j.jpag.2016.08.003. Epub 2016 Aug 22. PMID 27561981
- [Background] Espey E, Ogburn T, Leeman L, Singh R, Ostrom K, Schrader R. Effect of progestin compared with combined oral contraceptive pills on lactation: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):5-13. doi: 10.1097/AOG.0b013e31823dc015. PMID 22143258
- [Background] Acog.org. (2018). Medicaid Reimbursement for Postpartum LARC by State - ACOG. [online] Available at: https://www.acog.org/About-ACOG/ACOG-Departments/Long-Acting-Reversible-Contraception/Immediate-Postpartum-LARC-Medicaid-Reimbursement?IsMobileSet=false [Accessed 12 Jan. 2019].
- [Background] Ireland LD, Goyal V, Raker CA, Murray A, Allen RH. The effect of immediate postpartum compared to delayed postpartum and interval etonogestrel contraceptive implant insertion on removal rates for bleeding. Contraception. 2014 Sep;90(3):253-8. doi: 10.1016/j.contraception.2014.05.010. Epub 2014 May 24. PMID 24973904
- [Background] Phemister DA, Laurent S, Harrison FN Jr. Use of Norplant contraceptive implants in the immediate postpartum period: safety and tolerance. Am J Obstet Gynecol. 1995 Jan;172(1 Pt 1):175-9. doi: 10.1016/0002-9378(95)90109-4. PMID 7847530
- [Background] Dobromilsky KC, Allen PL, Raymond SH, Maindiratta B. A prospective cohort study of early postpartum etonogestrel implant (Implanon(R)) use and its effect on duration of lochia. J Fam Plann Reprod Health Care. 2016 Jul;42(3):187-93. doi: 10.1136/jfprhc-2014-101081. Epub 2015 Nov 6. PMID 26545933
- [Background] Horibe M, Hane Y, Abe J, Matsui T, Kato Y, Ueda N, Sasaoka S, Motooka Y, Hatahira H, Hasegawa S, Kinosada Y, Hara H, Nakamura M. Contraceptives as possible risk factors for postpartum depression: A retrospective study of the food and drug administration adverse event reporting system, 2004-2015. Nurs Open. 2018 Jan 17;5(2):131-138. doi: 10.1002/nop2.121. eCollection 2018 Apr. PMID 29599988
- [Background] Roberts TA, Hansen S. Association of Hormonal Contraception with depression in the postpartum period. Contraception. 2017 Dec;96(6):446-452. doi: 10.1016/j.contraception.2017.08.010. Epub 2017 Sep 1. PMID 28867443
- [Background] Flore M, Chen XL, Bonney A, Mullan J, Dijkmans-Hadley B, Hodgkins A, Evans G, Frew H, Lloyd G. Patients' perspectives about why they have their contraceptive Implanon NXT device removed early. Aust Fam Physician. 2016 Oct;45(10):740-744. PMID 27695725
- [Background] SAFE-T Pocket Card: Suicide Assessment Five-Step Evaluation and Triage for Clinicians. SAMHSA
- [Background] Higgins JA, Sanders JN, Palta M, Turok DK. Women's Sexual Function, Satisfaction, and Perceptions After Starting Long-Acting Reversible Contraceptives. Obstet Gynecol. 2016 Nov;128(5):1143-1151. doi: 10.1097/AOG.0000000000001655. PMID 27741195
- [Background] Meston CM, Derogatis LR. Validated instruments for assessing female sexual function. J Sex Marital Ther. 2002;28 Suppl 1:155-64. doi: 10.1080/00926230252851276. PMID 11898697
- [Background] Sanders JN, Higgins JA, Adkins DE, Stoddard GJ, Gawron LM, Turok DK. The Impact of Sexual Satisfaction, Functioning, and Perceived Contraceptive Effects on Sex Life on IUD and Implant Continuation at 1 Year. Womens Health Issues. 2018 Sep-Oct;28(5):401-407. doi: 10.1016/j.whi.2018.06.003. Epub 2018 Aug 18. PMID 30131221
- [Background] Li R, Fein SB, Chen J, Grummer-Strawn LM. Why mothers stop breastfeeding: mothers' self-reported reasons for stopping during the first year. Pediatrics. 2008 Oct;122 Suppl 2:S69-76. doi: 10.1542/peds.2008-1315i. PMID 18829834
- [Background] Odom EC, Li R, Scanlon KS, Perrine CG, Grummer-Strawn L. Reasons for earlier than desired cessation of breastfeeding. Pediatrics. 2013 Mar;131(3):e726-32. doi: 10.1542/peds.2012-1295. Epub 2013 Feb 18. PMID 23420922

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Insertion Group | Standard Postpartum Insertion Group
Started | 78 | 72
Modified Intention to Treat | 69 | 57
Completed | 62 | 53
Not Completed | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Immediate Insertion Group, Per Protocol: Immediate insertion within first 24 hours after delivery ENG implant insertion Intervention.
- Standard Postpartum Insertion Group, Per Protocol: Insertion of the Etonogestrel implant 4-6 weeks postpartum (changed post hoc to at least 2 weeks postpartum)
- Total: Total of all reporting groups
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol | Total
Number analyzed (Participants) | 62 | 53 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (5.5) | 27.2 (5.3) | 27.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 53 | 115
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latina | 44 | 44 | 88
  American Indian or Alaska Native | 4 | 7 | 11
  Black or African American | 2 | 1 | 3
  White | 34 | 26 | 60
  Other | 15 | 15 | 30
Parity [Mean (Inter-Quartile Range); unit: Parity] | 2 [1 to 3] | 1 [1 to 2] | 2 [1 to 3]
Previously used implant [Count of Participants; unit: Participants] | 26 | 16 | 42
Previously breastfed [Count of Participants; unit: Participants] | 33 | 23 | 56
Planning to breastfeed more than 6 months [Count of Participants; unit: Participants] | 51 | 47 | 98
Delivery mode [Count of Participants; unit: Participants]
  Vaginal | 51 | 39 | 90
  Cesarean | 9 | 13 | 22
  Operative vaginal | 2 | 1 | 3
Epidural [Count of Participants; unit: Participants] | 43 | 35 | 78
Recruitment site [Count of Participants; unit: Participants]
  University of New Mexico | 50 | 45 | 95
  University of Utah | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Continuation of Breastfeeding at 8 Weeks Postpartum
Description: Using a questionnaire the investigators seek to compare continuation of lactation between women in the immediate versus standard group. This will be assessed by answering a question with a dichotomous scale of yes or no in the follow-up questionnaire administer at 2,4,8,12 and 24 weeks postpartum.
Time Frame: For the primary outcome will be the first eight weeks after delivery.
Measure: Count of Participants; unit: Participants
Groups:
- Immediate: Implant Placed Within 24 Hours Postpartum -- Modified Intention-to-treat; Immediate: Implant Placed Within 24 Hours Postpartum -- Per Protocol: Immediate insertion in the first 24 hours after delivery ENG implant insertion Intervention.
- Standard: Implant Placed at Least 2 Weeks Postpartum -- Modified Intention-to-treat; Standard: Implant Placed at Least 2 Weeks Postpartum -- Per Protocol: Changed from beginning of study from "4-6 weeks weeks postpartum" to at "least 2 weeks postpartum."
  This change was decided after completing data collection for the following reasons:
  1. to increase sample size in the per-protocol group;
  2. to align with biologic plausibility in exposure to exogenous hormones as the "at least 2-week" interval is sufficiently remote from lactogenesis;
  3. to be consistent with the American College of Obstetricians and Gynecologists recommendation for earlier intiation of postpartum visits.
Arm/Group | Immediate: Implant Placed Within 24 Hours Postpartum -- Modified Intention-to-treat | Standard: Implant Placed at Least 2 Weeks Postpartum -- Modified Intention-to-treat | Immediate: Implant Placed Within 24 Hours Postpartum -- Per Protocol | Standard: Implant Placed at Least 2 Weeks Postpartum -- Per Protocol
Number analyzed (Participants) | 69 | 57 | 62 | 53
Participants | 54 | 45 | 48 | 43
Statistical Analysis 1: Comparison: Immediate: Implant Placed Within 24 Hours Postpartum -- Per Protocol vs Standard: Implant Placed at Least 2 Weeks Postpartum -- Per Protocol; To achieve 80% power with a 1-sided type 1 error of 5% utilizing the Z-test (unpooled), 62 participants would be required in each group, for a total of 124 participants. Accounting for expected loss to follow-up of 20%, we aimed to recruit 149 participants and rounded up to final recruitment goal of 150; Test type: Non-Inferiority — We used a 15% difference in our primary outcome for the non-inferiority margin as this is the upper end of the estimated prevalence of lactation failure in the literature and is consistent with previous studies (Neifert 2001, Gurtcheff 2011, Turok 2017); Risk Difference (RD) = 3.7, 95% CI 1-sided [lower limit -16.7]; The risk-difference between immediate and standard placement in the modified intention-to-treat analysis (mITT) was -0.6% with a -12.8% lower limit of the 95% confidence interval. In the mITT analysis, 78.3% (54/69) and 78.9% (45/57) of participants were breastfeeding at 8 weeks in the immediate and delayed groups, respectively

2. Secondary Outcome: Exclusive Breastfeeding
Description: Using a questionnaire the investigators seek to compare exclusive breastfeeding through 6 months postpartum between the immediate versus the standard group. This will be assessed by answering a trichotomous question with the following statement:
  If you are currently breastfeeding, are you:
  * Exclusively breastfeeding
  * Breastfeeding and supplementing breastfeeding with bottles of breast milk
  * Breastfeeding and supplementing breastfeeding with bottles of formula
Time Frame: Up to 24 weeks postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 56 | 53
Participants | 13 | 9

3. Secondary Outcome: Factors Associated With Breastfeeding Discontinuation.
Description: Using a questionnaire the investigators seek to compare factors associated with discontinuing breastfeeding between the immediate versus the standard group.
  Subjects were asked to rate the importance of seven different factors independently, on a 4-item Likert scale from 0 = Not at all important, to 3 = Very important
Time Frame: Up to 24 weeks postpartum.
Population: Some subjects provided partial data or no data at all.
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 28 | 26
score on a Likert scale
  Baby had trouble sucking or latching: number analyzed (Participants) | 28 | 25
  Baby had trouble sucking or latching | 0.5 [0 to 2.75] | 3 [0 to 3]
  Baby got sick | 0 [0 to 0] | 0 [0 to 0.25]
  I was sick | 0 [0 to 0] | 0 [0 to 2]
  Provider said baby was underweight | 0 [0 to 0] | 0 [0 to 1.25]
  Insufficient milk | 2 [0 to 3] | 2 [0 to 3]
  I had trouble; breast issues | 0 [0 to 0] | 1.5 [0 to 3]
  I quit breastfeeding; life issues | 2 [0 to 2] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Baby had trouble sucking or latching; Test type: Other; p = 0.221, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Baby got sick; Test type: Other; p = 0.786, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; I was sick; Test type: Other; p = 0.064, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Provider said baby was underweight; Test type: Other; p = 0.044, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Insufficient milk; Test type: Other; p = 0.666, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; I had trouble; breast issues; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; I quit breastfeeding; life issues; Test type: Other; p = 0.476, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Satisfaction With Postpartum Contraception Counseling
Description: Person-Centered Contraceptive Counseling Measure (PCCC Measure) pcccmeasure.ucsf.edu
  Scale range:
  1. Poor
  2. Fair
  3. Good
  4. Very Good
  5. Excellent
  Higher values represent higher satisfaction and patient-centeredness
Time Frame: At enrollment.
Population: Some subjects provided partial data or no data at all.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 62 | 53
score on a scale
  Respecting me as a person: number analyzed (Participants) | 61 | 41
  Respecting me as a person | 5 [5 to 5] | 5 [5 to 5]
  Letting me say what mattered to me about my birth control method: number analyzed (Participants) | 61 | 40
  Letting me say what mattered to me about my birth control method | 5 [4 to 5] | 5 [4 to 5]
  Taking my preferences about my birth control seriously: number analyzed (Participants) | 60 | 41
  Taking my preferences about my birth control seriously | 5 [4 to 5] | 5 [5 to 5]
  Giving me enough information to make the best decision about my birth control method: number analyzed (Participants) | 61 | 40
  Giving me enough information to make the best decision about my birth control method | 5 [5 to 5] | 5 [4 to 5]
Statistical Analysis 1: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Respecting me as a person; Test type: Other; p = 0.717, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Letting me say what mattered to me about my birth control method; Test type: Other; p = 0.808, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Taking my preferences about my birth control seriously; Test type: Other; p = 0.967, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Giving me enough information to make the best decision about my birth control method; Test type: Other; p = 0.826, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Postpartum Mood
Description: To compare postpartum mood as measured by Edinburgh Postnatal Depression Scale (EPDS) score at 2, 4, and 8 weeks postpartum. Results reported as a total score ranging from 0-30, no subscale scores. A higher scale represents a worse outcome, ie. is more predictive of a depressive disorder including postpartum depression.
Time Frame: At 2, 4, and 8 weeks postpartum.
Population: Some subjects provided partial data or no data at all.
Measure: Median (Inter-Quartile Range); unit: EPDS Score
Groups:
- Standard Postpartum Insertion Group, Per Protocol: Insertion of the Etonogestrel implant 4-6 weeks postpartum (changed post hoc to at least 2 weeks postpartum
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 62 | 53
EPDS Score
  2 weeks postpartum: number analyzed (Participants) | 25 | 20
  2 weeks postpartum | 2 [1 to 5] | 1 [1 to 8]
  4 weeks postpartum: number analyzed (Participants) | 25 | 17
  4 weeks postpartum | 2 [1 to 6] | 4 [1 to 7]
  8 weeks postpartum: number analyzed (Participants) | 23 | 18
  8 weeks postpartum | 3 [1 to 6] | 4 [1 to 7]
Statistical Analysis 1: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 2 weeks postpartum; Test type: Other; p = 0.264, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 4 weeks postpartum; Test type: Other; p = 0.414, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 8 weeks postpartum; Test type: Other; p = 0.482, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Sexual Function
Description: To compare postpartum sexual function as measured by Female Sexual Function Index (FSFI) score. Minimum score 2, Maximum score 36. Subscales are combined by first totaling the scores for the individual questions in that domain (ex. for Desire, the sum of scores for questions 1 and 2). That total is then multiplied by the factor for that domain, which is listed in the table above. The output is the final score for that domain, and will fall within the minimum and maximum scores listed in the table above.
  For every domain, a lower score indicates either no sexual activity or negative outcomes in that domain, while a higher score indicates positive outcomes in that domain.
Time Frame: At 4, 8, and 12 weeks postpartum
Population: Some subjects provided partial data or no data at all.
Measure: Median (Inter-Quartile Range); unit: FSFI Score
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 62 | 53
FSFI Score
  4 weeks postpartum: number analyzed (Participants) | 43 | 30
  4 weeks postpartum | 6 [4.4 to 19.5] | 6 [3.9 to 7.7]
  8 weeks postpartum: number analyzed (Participants) | 43 | 38
  8 weeks postpartum | 16 [4.8 to 25.4] | 18.5 [8 to 29.3]
  12 weeks postpartum: number analyzed (Participants) | 38 | 36
  12 weeks postpartum | 19.9 [7 to 27.9] | 21.9 [8.6 to 28.2]
Statistical Analysis 1: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 4 weeks postpartum; Test type: Other; p = 0.583, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 8 weeks postpartum; Test type: Other; p = 0.062, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 12 weeks postpartum; Test type: Other; p = 0.705, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Postpartum Bleeding Days
Description: To compare the total number of days of postpartum bleeding in the immediate versus standard group.
  This is a secondary outcome for which analysis is ongoing.
Time Frame: At 2, 4, and 8 weeks postpartum.
Population: Some subjects provided partial data: i.e. only provided responses for some days or no data at all.
Measure: Median (Inter-Quartile Range); unit: Days with bleeding
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 62 | 53
Days with bleeding
  2 weeks postpartum: number analyzed (Participants) | 33 | 22
  2 weeks postpartum | 14 [14 to 14] | 14 [14 to 14]
  4 weeks postpartum: number analyzed (Participants) | 31 | 23
  4 weeks postpartum | 14 [14 to 14] | 12 [7 to 14]
  8 weeks postpartum: number analyzed (Participants) | 29 | 31
  8 weeks postpartum | 25 [0 to 28] | 11 [1 to 28]
Statistical Analysis 1: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 2 weeks postpartum; Test type: Other; p = 0.60, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 4 weeks postpartum; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; 8 weeks postpartum; Test type: Other; p = 0.36, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Satisfaction With the ENG Implant
Description: Using a questionnaire the investigators seek to compare participant satisfaction with the ENG implant between the immediate versus the standard group.
  Scale: 0= Unsatisfied, 1=Satisfied, 2=Very satisfied
Time Frame: At 8 weeks postpartum
Population: Some subjects provided partial data or no data at all.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 36 | 20
score on a scale | 1 [1 to 1] | 1 [1 to 2]
Statistical Analysis 1: Comparison: Immediate Insertion Group, Per Protocol vs Standard Postpartum Insertion Group, Per Protocol; Test type: Other; p = 0.0376, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Timing of Breastfeeding Discontinuation Through 24 Weeks Postpartum Between Immediate and Standard Groups.
Description: To compare timing of breastfeeding discontinuation through 6 months postpartum between the immediate versus the standard group.
Time Frame: Up to 24 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Insertion Group, Per Protocol | Standard Postpartum Insertion Group, Per Protocol
Number analyzed (Participants) | 51 | 48
Participants | 24 | 24

ADVERSE EVENTS:
Time Frame: 5 years
Description: The all-cause mortality event reported below was discovered during chart review. At that point in time, study recruitment and all prospective data collection from participants had already concluded. The IRB was notified, reviewed the case, and concluded that this death was unrelated to study participation, and therefore did not increase the overall risk of harm from participation.
Arm/Group | Immediate Insertion Group | Standard Postpartum Insertion Group
All-Cause Mortality (participants affected / at risk) | 0/78 | 1/72
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/72
Other Adverse Events (participants affected / at risk) | 0/78 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03978598/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03978598/ICF_002.pdf